CLINICAL TRIAL: NCT05941195
Title: Investigation of the Effect of Cognitive Behavioral Approach-Based Psychoeducation on Addiction Profile, Self-efficacy and Addiction Course in Substance Use Disorder Randomized Controlled Experimental Study
Brief Title: Investigation of the Effect of Cognitive Behavioral Approach-Based Psychoeducation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Cihan Kocairi, Research Assistant, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Adnan MU
Record Dates: First submitted 2023-06-02; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Substance Use Disorders; Self Efficacy; Addiction
Keywords: Substance Use Disorder; Psychosocial Intervention; Self Efficacy; Psychiatric Nursing
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: Following recruitment, person who the substance use disorder were divided into a study and a control group by randomization (1:1 randomization)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- psychoeducation applied experimental group (Experimental): The patients in the experimental group received a total of 5 weeks (9 sessions) of cognitive-behavioral-based psychoeducation, consisting of 45-60 minutes, 2 sessions per week and the first session preparation session. In the sessions, the topics determined by using learning activities such as lecture, discussion, summarization, role-play, question/answer and exercises were explained and discussed. At the end of each session, homework was given to facilitate the patient's cognitive and behavioral change between sessions.
  Interventions: Other: Psychoeducation
- non-intervention control group (No Intervention): Control group: The control group continued to receive the routine care.

INTERVENTIONS:
Other: Psychoeducation — In the cognitive behavioral approach based psychoeducation given to the experimental group patients; "Addiction and Its Effects", "Increasing and Maintaining Motivation", "The Cognitive Model and the Cognitive Model of Addiction", "Automatic Thoughts That Increase Impulse to Substance Use", "Dysfunctional Beliefs Regarding Substance Use", "High Risk Situations and Coping Skills", " The topics of "Prevention of Slippage and Recurrence" and "Problem Solving" are included.
  Arms: psychoeducation applied experimental group

SUMMARY:
This study, which was planned to examine the effects of cognitive behavioral approach-based psychoeducation on addiction profiles, self-efficacy levels and addiction courses in patients with substance use disorders, was carried out as a randomized controlled experimental study.

DETAILED DESCRIPTION:
It can be said that alcohol/substance nurses, by applying cognitive behavioral approach-based psychoeducation to patients with substance use disorders, can have a positive effect on reducing the severity of addiction, increasing their self-efficacy levels, and providing the care, education and counseling support that patients need.

The aim of this study is to examine the effects of cognitive behavioral approach-based psychoeducation applied to patients with substance use disorder on addiction profiles, self-efficacy levels and addiction courses.

ELIGIBILITY:
Inclusion Criteria:

1. To be diagnosed with "Substance Use Disorder" according to The Diagnostic and Statistical Manual of Mental Disorders-V,
2. To be over 18 years old,
3. Volunteering to participate in the research.

Exclusion Criteria:

1. Other than Substance Use Disorder, chronic, requiring ongoing help and care the presence of a medical illness,
2. Being illiterate (the types of scales to be used must be self-report forms) because of).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Addiction Profile Index (Bapi) Clinical Form | The first measurement was made in the 1st week.
  Addiction Profile Index Clinical Form was created by adding 21 questions to the Addiction Profile Index developed in 2012 to measure the severity of addiction. It consists of 58 questions in total and has 11 sub-dimensions. It evaluates different dimensions of addictions of alcohol and substance users. Two of the six domains of the scale measure mental state, while the others measure some personal characteristics related to addiction .
Addiction Profile Index (Bapi) Clinical Form | The last measurement was made at the 5th week.
  Addiction Profile Index Clinical Form was created by adding 21 questions to the Addiction Profile Index developed in 2012 to measure the severity of addiction. It consists of 58 questions in total and has 11 sub-dimensions. It evaluates different dimensions of addictions of alcohol and substance users. Two of the six domains of the scale measure mental state, while the others measure some personal characteristics related to addiction.
Addiction Outcome Assessment Index (AOAI) | The first measurement was made in the 1st week.
  The Addiction Outcome Index (BASI) was developed to measure the treatment course and recovery level of addiction in all areas and to be used in follow-up. The score that can be obtained from the scale is between 0-32. A decrease of 3.5 points from the total score of the scale in clinical follow-up indicates a reliable change .
Addiction Outcome Assessment Index (AOAI) | The last measurement was made at the 5th week.
  The Addiction Outcome Index (BASI) was developed to measure the treatment course and recovery level of addiction in all areas and to be used in follow-up. The score that can be obtained from the scale is between 0-32. A decrease of 3.5 points from the total score of the scale in clinical follow-up indicates a reliable change .
Self-Efficacy Scale (SES) | The first measurement was made in the 1st week.
  The scale was first developed in the English language in 1982. It was adapted into Turkish in 1999 and follows the course of self-efficacy expectations that need to be changed in individual therapy during the therapy process. The Self-Efficacy Scale consists of 23 items and 4 sub-factors. A minimum of 23 and a maximum of 115 points can be obtained from the scale. A high total score from the scale indicates that the individual's self-efficacy perception is at a good level.
Self-Efficacy Scale (SES) | The last measurement was made at the 5th week.
  The scale was first developed in the English language in 1982 . It was adapted into Turkish in 1999 and follows the course of self-efficacy expectations that need to be changed in individual therapy during the therapy process. The Self-Efficacy Scale consists of 23 items and 4 sub-factors. A minimum of 23 and a maximum of 115 points can be obtained from the scale. A high total score from the scale indicates that the individual's self-efficacy perception is at a good level.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma DEMİRKIRAN, Phd, Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Aydın Adnan Menderes University Faculy of Nursing, Division Mental HealthNursing, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request
Supporting Information: CSR
Time Frame: 2 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.

REFERENCES:
- [Background] Ögel K, Koç C, Başabak A, İşmen EM, Görücü S. Bağımlılık profil indeksi klinik formunun (BAPİ-K) geliştirilmesi: Geçerlik ve güvenilirlik Çalışması. Bağımlılık Dergisi.2015; 16(2), 57-69.
- [Background] Simsek M, Dinc M, Ogel K. The Validity aand Reliability of the Addiction Outcome Assessment Index (AOAI). Turk Psikiyatri Derg. 2021 Summer;32(2):129-136. doi: 10.5080/u23461. English, Turkish. PMID 34392509
- [Background] Sherer M, Maddux JE, Mercandante B, Prentice-Dunn S, Jacobs B, Rogers R W. The self-efficacy scale: Construction and validation. Psychological reports.1982; 51(2), 663-671.
- [Background] Gözüm S, Aksayan S. Öz-etkililik-yeterlik ölçeği'nin türkçe formunun güvenilirlik ve geçerliliği. Anadolu Hemşirelik ve Sağlık Bilimleri Dergisi. 1999; 2(1): 21-34.